CLINICAL TRIAL: NCT06365411
Title: GEnomic Medicine in Kidney Transplantation Study
Acronym: GEM-KiT
Status: Not yet recruiting | Type: Observational
Sponsor: Western Sydney Local Health District (Other)
Responsible Party: Principal Investigator, Jennifer Li, Nephrologist and Transplant Physician, Western Sydney Local Health District
Other Study IDs: GEM-KiT
Record Dates: First submitted 2024-03-10; First posted 2024-04-15 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-04

CONDITIONS: Transplant Complication; Kidney Transplant Rejection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sampling: all patients will submit blood samples (approximately 10 teaspoons), including
  * Blood (15ml) drawn into PAX gene tubes for extraction of genomic material (eg DNA, RNA)
  * Kidney biopsy sample: For patients undergoing kidney biopsy procedure for any clinical indication (part of their clinical care, independent of the study), a dedicated sample of kidney biopsy may be collected for the study with the patient's permission
  * Mid-stream urine sample for pellet and supernatant and then stored at -80'c
  * Faecal sample in dedicated gut microbiome kits and then stored at -80'c
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Kidney Transplant Recipients: Enrolled at time of transplant or post transplant
  Interventions: Diagnostic Test: Biomarker discovery and validation - with focus on genomic biomarkers

INTERVENTIONS:
Diagnostic Test: Biomarker discovery and validation - with focus on genomic biomarkers — Biomarker discovery and validation - with focus on genomic biomarkers

SUMMARY:
Investigator led, prospective, observational cohort study to detect genomic features which can predict outcomes following kidney transplantation.

1. Determine non-HLA genomic mismatches between donor-recipient pairs which impact kidney allograft survival following transplantation
2. Derive polygenic risk scores on pre-transplant blood and/or kidney biopsy samples which predict kidney allograft dysfunction
3. Derive polygenic risk scores on post-transplant blood and/or kidney biopsy samples which predict kidney allograft dysfunction

ELIGIBILITY:
Inclusion Criteria: All participants included in the study must be age ≥ 18 years old at time of enrolment and

1. able to provide informed consent (interpreter permitted) for enrolment
2. consenting to longitudinal follow up (can withdraw post enrolment)
3. consenting to provide samples for biobanking, including blood, urine, faecal and/or kidney biopsy tissue (collected prospectively, separate to routine care)

Exclusion Criteria: Patients will be excluded from the study if they are

1. unable (or unwilling) to provide consent, or
2. have life-expectancy less than 6-months, or
3. have received a haematopoietic stem cell transplant in the past 5 years.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult, kidney transplant (or kidney-pancreas transplant) recipients
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-06-03 (Estimated); Primary Completion 2030-01-01 (Estimated); Study Completion 2035-01-01 (Estimated)

PRIMARY OUTCOMES:
Death censored graft loss (DCGL) | At biopsy or during study follow up after biopsy (expected average over 60-months)
  Loss of functioning kidney transplant (not counted if patient died with functioning graft)
Biopsy proven rejection (BPAR) | At biopsy or during study follow up after biopsy (expected average 12-months)
  Rejection diagnosed on kidney transplant biopsy

SECONDARY OUTCOMES:
All cause graft loss | At biopsy or during study follow up after biopsy (expected average over 60-months)
  DCGL or death with functioning graft
Death | Any time during or after biopsy (expected over 60-months)
  Death
Treatment resistant rejection | At biopsy or during study follow up after biopsy (expected average 12-months)
  Persistent rejection despite additional glucocorticoids and/or upscaling of maintenance immunosuppression
Hospital admission or emergency attendance | At biopsy or during study follow up after biopsy (expected average 12-months)
  Hospital admission or emergency department visit for any reason
Delayed Graft Function (DGF) | within the first 7 days post transplantation
  Need for dialysis within the first 7 days post transplantation
Kidney function | Months 1, 3, 12, 24, 36, 48, 60, 120 post transplantation
  serum creatinine and eGFR post transplantation
Albuminuria | Months 1, 3, 12 any time after 12-months trnasplantation
  albumin in the urine (UACR)
Surrogate end-point markers | Months 3, 12, 24, 36, 48 and 60, 120 post transplantation
  eGFR slope and iBOX scores
Borderline rejeciton | At biopsy or during study follow up after biopsy (expected average 12-months)
  Based on banff scoring criteria for kidney biospies
chronic rejection; chronic transplant glomerulopathy; and interstitial fibrosis and tubular atrophy (IFTA) scores | At biopsy or during study follow up after biopsy (expected average over 12-months)
  Based on banff scoring for kidney biopsies
Recurrent disease | At biopsy or during study follow up after biopsy (expected average 60-months)
  recurrence of original disease causing kidney failure
BK virus complications | At biopsy or during study follow up after biopsy (expected average 12-months)
  Viremia or virus associated nephropathy
Major cardiovascular complications | At biopsy or during study follow up after biopsy (expected average 60-months)
  3-point MACE: non fatal stroke, non fatal myocardial infarction, cardiovascular death
Major infectious complications | At biopsy or during study follow up after biopsy (expected average 60-months)
  any major fungal, bacterial or viral infection
Malignancy post transplantation | At biopsy or during study follow up after biopsy (expected average 60-months)
  any cancer type
Kidney biopsy transcriptomic signature | At biopsy - based on collected tissue sample
  Based on bulk and/or spatial transcriptomic experiments
Kidney cell type composition | At biopsy - based on collected tissue sample
  Cell type phenotyping of immune and kidney cell types
Proteinomic signature | At biopsy or during study follow up after biopsy (expected average 12-months)
  mass spectrometry or spatial proteinomic results

IPD SHARING:
Plan to Share IPD: No